CLINICAL TRIAL: NCT03884608
Title: BIO-LIBRA Clinical Study
Brief Title: Analysis of Both Sex and Device Specific Factors on Outcomes in Patients with Non-Ischemic Cardiomyopathy
Acronym: BIO-LIBRA
Status: Completed | Type: Observational
Sponsor: Biotronik, Inc. (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: BIO-LIBRA
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cardiomyopathies; Gender; Implantable Defibrillator User
MeSH Terms: conditions — Cardiomyopathies; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this registry is to prospectively assess outcomes of device-treated ventricular tachyarrhythmias and all-cause mortality in non-ischemic cardiomyopathy patients indicated for ICD or CRT-D implantation for the primary prevention of sudden cardiac death. Differences in outcomes will be evaluated by sex and by device type.

DETAILED DESCRIPTION:
The BIO-LIBRA Study will gather information about women and men with non-ischemic cardiomyopathy who are treated with implanted ICD and CRT-D devices from many locations across the United States. The BIO-LIBRA Study will look at the results of treatment in women and men enrollees. The two primary goals are: 1) to learn if there are differences in treatment response based on the patient's sex; and 2) to learn if there are differences in patient outcomes based on device type.

There is a special focus on women in the BIO-LIBRA Study. Usually, only about 25% of people in prior device studies have been women. Yet heart disease is the number-one cause of death for women - one in three deaths each year. The BIO-LIBRA Study would like to have a more balanced study which includes more women than in prior studies. The goal is for at least 40% of the people participating in the study to be women.

The study will observe up to 1,000 women and men over a three-year period following the device implant. Utilizing information collected at annual doctor visits and scheduled transmission reports from the implanted device in between these visits, the BIO-LIBRA Study will be able to evaluate some of the common risks of non-ischemic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets current guideline-defined indication for de novo, primary prevention ICD or CRT-D implantation
2. Patient has non-ischemic etiology of cardiomyopathy
3. Patient is successfully implanted with a de novo BIOTRONIK ICD or CRT-D device and commercially available leads no more than 30 days prior to consent or is scheduled for de novo implantation of a BIOTRONIK ICD or CRT-D device no more than 30 days post consent
4. Patient is able to understand the nature of the study and provide informed consent
5. Patient is available for standard of care follow-up visits to occur at least yearly at the study site for to the expected 3 years of follow-up
6. Patient is willing to utilize BIOTRONIK Home Monitoring® via CardioMessenger
7. Patient age is greater than or equal to 18 years

Exclusion Criteria:

1. Patient meets secondary prevention ICD indication
2. Patient has ischemic etiology of cardiomyopathy
3. Patient is enrolled in any investigational cardiac device or drug trial that might significantly affect the studied outcomes
4. Patient is expected to receive heart transplantation or ventricular assist device within 1 year
5. Patient life expectancy is less than 1 year
6. Patient reports pregnancy at the time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients selected for participation should be from the investigator's general patient population according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Evaluation of the combined risk of all-cause mortality and treated ventricular tachycardia (VT) or ventricular fibrillation (VF) events | 3 years post-implant
  Evaluate the combined risk of all-cause mortality and treated ventricular tachycardia (VT) or ventricular fibrillation (VF) events by sex and by implanted device type

SECONDARY OUTCOMES:
Rate of all-cause mortality | 3 years post-implant
  Rate of all-cause mortality will be analyzed for the total cohort, as well as by sex and by the implanted device type
Rate of treated ventricular tachycardia (VT) or ventricular fibrillation (VF) events | 3 years post-implant
  Rate of treated ventricular tachycardia (VT) or ventricular fibrillation (VF) events will be analyzed for the total cohort, as well as by sex and by the implanted device type
Rate of cardiac death | 3 years post-implant
  Rate of cardiac death will be analyzed for the total cohort, as well as by sex and by the implanted device type
Rate of sudden cardiac death | 3 years post-implant
  Rate of sudden cardiac death will be analyzed for the total cohort, as well as by sex and by the implanted device type
Comparison of the Seattle Proportional Risk Model (SPRM) predicted incidence of sudden death to the observed incidence of death | 3 years post-implant
  Comparison of the Seattle Proportional Risk Model (SPRM) predicted incidence of sudden death to the observed incidence in this patient population

OTHER OUTCOMES:
Evaluation of cardiovascular and diabetes medication use and dosage during the study | 3 years post-implant
  Evaluation of cardiovascular and diabetes medication use and dosage during the study in both ICD and CRT-D patients stratified by sex
Assessment of left ventricular reverse remodeling by echocardiography at 12 months for CRT-D patients | 12 months post-implant
  Assessment of left ventricular reverse remodeling using echocardiography at 12 months for patients implanted with CRT-D as characterized by the change compared to the baseline assessment of the left ventricular ejection fraction (LVEF) and left ventricular end-systolic volume (LVESV)
Rate of inappropriate ICD therapy | 3 years post-implant
  Analysis of the rate of inappropriate ICD therapy (ICD delivered ATP or shock for rhythms other than VT/VF) in both ICD and CRT-D patients stratified by sex
Rate of ventricular tachycardia (VT) or ventricular fibrillation (VF) events treated with shock only | 3 years post-implant
  Analysis of the rate of ventricular tachycardia (VT) or ventricular fibrillation (VF) events treated with shock only by sex and by device type
Rate of observed major complications | 3 years post-implant
  Evaluation of the observed major complication rates, including the overall rate and rates of individual major complications in both ICD and CRT-D patients stratified by sex

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Kutyifa, MD, PhD, Principal Investigator — University of Rochester; Jeanne Poole, MD, Principal Investigator — University of Washington
Locations (49):
- United States (49):
  - Southview Cardiovascular Associates, Birmingham, Alabama
  - Cardiology Associates of Mobile, Fairhope, Alabama
  - Eisenhower Desert Cardiology, Rancho Mirage, California
  - UC Davis Medical Center, Sacramento, California
  - Cardiology Associates Medical Group, Ventura, California
  - Cardiovascular Institute of North Colorado, Greeley, Colorado
  - University of Florida, Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health, Inc., Orlando, Florida
  - BayCare Medical Group Cardiology, Safety Harbor, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Saint Alphonsus Heart Care, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Traverse Heart and Vascular, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Cardiology Associates Research, Tupelo, Mississippi
  - Mercy Clinic Heart and Vascular, St Louis, Missouri
  - Logan Health Research, Kalispell, Montana
  - NYP Brooklyn Methodist Hospital, Brooklyn, New York
  - Trinity Medical WNY, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Sanger Heart and Vascular, Charlotte, North Carolina
  - East Carolina University Physicians, Greenville, North Carolina
  - Heart Rhythm Associates, Greenville, North Carolina
  - Cape Fear Heart Associates, Wilmington, North Carolina
  - Novant Health Winston Salem Cardiology, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - ProMedica Physicians Cardiology, Toledo, Ohio
  - Penn State Health Milton S Hershey, Hershey, Pennsylvania
  - Geisinger Heart and Vascular Center, Scranton, Pennsylvania
  - Upstate Cardiology, Greenville, South Carolina
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Carolina Arrhythmia Consultants, Mt. Pleasant, South Carolina
  - Cardiology Consultants, Spartanburg, South Carolina
  - University of Tennessee Erlanger Cardiology, Chattanooga, Tennessee
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant level data collected within the study will be shared for approved requests of subsidiary studies not specifically pre-planned within the protocol.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available beginning no later than 12 months and ending no earlier than 3 years following publication.
Access Criteria: Proposals should be directed to BIOTRONIK Clinical Studies (BIOTRONIK Inc., Attn: Clinical Studies, 6024 Jean Road, Lake Oswego, OR; 1-800-547-0394). The Principal Investigator and Co-Principal Investigator, in consultation with BIOTRONIK, will review and critique subsidiary requests for scientific merit, fiscal feasibility, and logistical feasibility. They will additionally consider if the proposed publication fits into the overall BIO-LIBRA publication plan. If approved, the data requestors will need to sign a data use/access agreement prior to obtaining the data and agree to have the Principal Investigator and Co-Principal Investigator as co-authors.

REFERENCES:
- [Derived] Kutyifa V, Di Biase L, Prasad KV, Torres V, Hesselson A, McCotter CJ, Harris G, Cox K, Schleede S, Heist EK, McNitt S, Brown MW, Miller C, Beck CA, Poole J; BIO-LIBRA Investigators. Contemporary medical therapy, sex-specific characteristics, and outcomes of patients with non-ischemic cardiomyopathy: a prespecified interim analysis of the BIO-LIBRA study. EClinicalMedicine. 2025 Jul 13;86:103337. doi: 10.1016/j.eclinm.2025.103337. eCollection 2025 Aug. PMID 40697957